CLINICAL TRIAL: NCT05048030
Title: Survey of Lifestyle and Its Feelings in Families of Patients in Home Parenteral Nutrition
Acronym: NPAD
Status: Completed | Type: Observational
Sponsor: Imagine Institute (Other)
Collaborators: Hôpital Necker-Enfants Malades (Other)
Responsible Party: Sponsor
Other Study IDs: HJ-21-NPAD
Record Dates: First submitted 2021-09-01; First posted 2021-09-17 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Home Parenteral Nutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Description of the life style of patients and families during the course of long term HPN.

1. Evaluation of the familial impact of HPN, and the way it is perceived
2. Evaluation of the satisfaction regarding the management by the multi-professional team (Medical, nursing, home care company and logistic, social, psychologist etc..) for improving the global management of these challenging patients
3. Analysis of the factors related to specific distress and the protective factors

DETAILED DESCRIPTION:
Gastrointestinal diseases may cause intestinal failure (IF) requiring long term parenteral nutrition (PN) which is, most of the time, performed at home (HPN).

However such conditions represent a great burden for the parents and the family.

The birth of a child with such disease changes the life of the entire family including life style, leisures, social relationships and professional activities.

These condition obligate to change the personal and familial organization according to the course of the disease. The PN treatment which was seen as life saving when first started might become a burden altogether physically and psychologically for the child and his/her family.

The Necker-Enfants Malades hospital developed home PN in the early eighties as an alternative to very long hospitalizations.

Nowadays, there are 7 expert centers for HPN in France. The Necker HPN program is the oldest and the largest looking after i a third of the 400 children on HPN in France.

Our organization is based on a specializednursing team together with medical doctors specialized in pediatric clinical nutrition.

The nursing team is also a teaching team for training the parents for daily PN care. The HPN team works in collaboration with professional partners: pharmacists, dieticians, psychologists, occupational therapistsand speech specialists as well as with social workers.

Results of our clinical activities have been published in international peer review journals. However those publications reported only clinical data in terms of diagnosis, prognosis, mortality, morbidity and growth.There was any data on family quality of life (QOL) and on life style changes (LSC). In other words, by reporting only on medical aspects, there was any analyze on familial, psychosocial and professional impact of long term HPN.

ELIGIBILITY:
Inclusion Criteria:

* Patients followed up by the Necker HPN expert center
* HPN ≥ 12 months
* HPN between 2004 and 2020
* Parents reading and writing French language

Exclusion Criteria:

* Refusal of the parents to participate to the survey

Ages: 18 Months to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children, and their entire family, with gastrointestinal diseases and intestinal failure (IF) requiring long term parenteral nutrition, performed at home (HPN).
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Demographic data and socio-familial life style with a child on long-term | Base line
  socio-familial life style
Data involving the management of HPN | Base line
  Logistics organization

SECONDARY OUTCOMES:
Perception of the familial impact of HPN on life style in case of protracted HPN dependency | Base line
  Child development
Satisfaction level of the management by the HPN expert center | Base Line
  Medical and nursing logistics
Factors influencing the familial burden | Base Line
  Type of disease

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Goulet, MD, PHD, Study Director — Department of Pediatric Gastroenterology-Hepatology-Nutrition, National Reference Center for Rare Digestive Diseases, Pediatric Intestinal Failure Rehabilitation Center
Locations (1):
- Hopital Necker - Enfants malades, Paris, France